CLINICAL TRIAL: NCT04482907
Title: Randomized Placebo Controlled Clinical Study of Anethum Graveolens L. (Dill) in Thyroiditis and Nodular Goiter Patients
Brief Title: Effect of Dill in Thyroiditis and Nodular Goiter Patients
Acronym: Dill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12.2014/21
Record Dates: First submitted 2020-07-16; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Nodule
Keywords: Anethum graveolens L.; Thyroiditis; Nodular Goiter
MeSH Terms: conditions — Thyroid Nodule; Thyroiditis; Goiter, Nodular

STUDY DESIGN:
Intervention Model Description: Two groups were created. Patients with thyroid nodules were divided into two groups given dill and placebo. The study was planned for 90 days. 900 mg of powder dill was given daily to the dill group. Placebo was given to the control group. Serum thyroid stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), anti-thyroid peroxidase (anti-TPO), anti-thyroglobulin (Anti-Tg) and C-reactive protein (CRP) levels of both groups were examined at the beginning and at the end of the study. Thyroid nodule dimensions were measured at the beginning and at the end of the study by ultrasonography. The results were evaluated statistically.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving dill (Active Comparator): They took 3 meals a day, 3x300 mg dry dill powder by mouth. They bought dry dill powder for 90 days.
  Interventions: Dietary Supplement: Giving dill by mouth capsule to the study group and placebo capsule by mouth to the control group.
- Group receiving placebo (Placebo Comparator): They took 3 meals a day and 3 cellulose placebo capsules by mouth. They took placebo capsules for 90 days.
  Interventions: Dietary Supplement: Giving dill by mouth capsule to the study group and placebo capsule by mouth to the control group.

INTERVENTIONS:
Dietary Supplement: Giving dill by mouth capsule to the study group and placebo capsule by mouth to the control group. — Tests from intravenous blood: TSH, fT3, fT4, anti-TPO, Anti-Tg, CRP
  Other Names: Taking blood from the arm intravenously at the beginning and end of the study and looking for thyroid hormones from this blood.

SUMMARY:
The aim of the study was to investigate the functional and morphological effects of Anethum graveolens L. in patients with thyroiditis and nodular goiter by evaluating hormone levels, anti-Inflammatory markers and comparing thyroid nodule sizes measured by ultrasonography for 90 days.

The effect of Anethum graveolens L. was evaluated in euthyroid goiter patients diagnosed with benign thyroid nodule via fine needle aspiration biopsy. Aerial parts of Anethum graveolens L. were dried and grinded to yield a fine powder. Size 1 hydroxypropyl methylcellulose capsules were filled with 300 mg powder. Placebo was prepared in the same manner using maltodextrin. Patients were suggested to take 3 pills a day. Blood samples were collected at the initial and the final day for thyroid stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), anti-thyroid peroxidase (anti-TPO), anti-thyroglobulin (Anti-Tg) and C-reactive protein (CRP) analysis. Nodule sizes were also measured at the beginning and at the end of the trial with ultrasonography to identify the changes and effectiveness of dill dosage forms.

After 90 days in the study, the status of TSH, fT3, fT4, anti-TPO and CRP levels were examined in the group with and without Anethum graveolens L..

Again, after the study, the size of thyroid nodules was evaluated in the group who received and did not receive Anethum graveolens L. by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* To have multi-nodular goiter,
* To be a benign result in fine needle aspiration biopsy,
* Euthyroid must be sick,
* Must be sick over the age of 18,
* To accept the research.

Exclusion Criteria:

* Thyroid function tests non-euthyroid individuals,
* To have a malignant result in thyroid biopsy,
* Not giving approval,
* To be renal failure,
* Benign pregnant,
* Taking blood thinning drugs

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Comparison of thyroid stimulating hormone (TSH) between groups | 90 days
  At the beginning and at the end of the study, the levels of serum TSH were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of free triiodothyronine (fT3) between groups | 90 days
  At the beginning and at the end of the study, the levels of serum fT3 were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of free thyroxine (fT4) between groups | 90 days
  At the beginning and at the end of the study, the levels of serum fT4 were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of anti-thyroid peroxidase (anti-TPO) between groups | 90 days
  At the beginning and at the end of the study, the levels of anti-TPO were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of anti-thyroglobulin (Anti-Tg) between groups | 90 days
  At the beginning and at the end of the study, the levels of serum Anti-Tg were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of C-reactive protein (CRP) between groups | 90 days
  At the beginning and at the end of the study, the levels of serum CRP were measured and statistically compared in groups given Anethum graveolens L. and placebo.
Comparison of ultrasound and thyroid nodule sizes between groups | 90 days
  At the beginning and end of the study, thyroid nodule sizes (mm) were measured and statistically compared in groups given Anethum graveolens L. and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegul Yabacı, research, Study Chair — Bezmialem Vakif University
Locations (1):
- Sabahattin Destek, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When published as a full article in a journal indexed, IPD will be shared.

REFERENCES:
- [Result] Jana S, Shekhawat GS. Anethum graveolens: An Indian traditional medicinal herb and spice. Pharmacogn Rev. 2010 Jul;4(8):179-84. doi: 10.4103/0973-7847.70915. PMID 22228959
- [Result] Orhan IE, Senol FS, Ozturk N, Celik SA, Pulur A, Kan Y. Phytochemical contents and enzyme inhibitory and antioxidant properties of Anethum graveolens L. (dill) samples cultivated under organic and conventional agricultural conditions. Food Chem Toxicol. 2013 Sep;59:96-103. doi: 10.1016/j.fct.2013.05.053. Epub 2013 Jun 10. PMID 23764360
- [Result] Antonelli A, Ferrari SM, Corrado A, Di Domenicantonio A, Fallahi P. Autoimmune thyroid disorders. Autoimmun Rev. 2015 Feb;14(2):174-80. doi: 10.1016/j.autrev.2014.10.016. Epub 2014 Oct 25. PMID 25461470
- [Result] Kratky J, Vitkova H, Bartakova J, Telicka Z, Antosova M, Limanova Z, Jiskra J. Thyroid nodules: pathophysiological insight on oncogenesis and novel diagnostic techniques. Physiol Res. 2014;63 Suppl 2(Suppl 2):S263-75. doi: 10.33549/physiolres.932818. PMID 24908232
- [Result] Yang ML, Lu B. Treatment of Goiter with Traditional Chinese Medicine Regimen Xing Qi Hua Ying Tang: A Clinical Study on 72 Patients with Multinodular and Diffuse Goiter. J Altern Complement Med. 2018 Apr;24(4):374-377. doi: 10.1089/acm.2017.0138. Epub 2017 Dec 7. PMID 29215302
- [Result] Altay M, Ates I, Kaplan Efe F, Karadag I. Does Use of Anethum Graveolens Affected Thyroid Hormone Levels and Thyroid Nodules? Am J Ther. 2017 Sep/Oct;24(5):e627-e629. doi: 10.1097/MJT.0000000000000511. No abstract available. PMID 27753646